CLINICAL TRIAL: NCT04910204
Title: Time Sensitivity of Adaptive Neuroplasticity and Functional Recovery Related to FEST in Combination with TST for Rehabilitation of Upper Extremity Function of Individuals with Tetraplegia
Brief Title: Time-effect of FEST+TST in the Upper-extremity Rehabilitation of Individuals with Traumatic SCI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Julio Furlan, MD, Neurologist, University Health Network, Toronto
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 19-6286
Record Dates: First submitted 2021-05-07; First posted 2021-06-02 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Spinal Cord Injuries
Keywords: functional electrical stimulation; task-specific training; upper limb rehabilitation
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early FEST + TST (Experimental): Participants will receive FEST+TST at 3 to 6 months from SCI onset.
  Interventions: Other: FES Therapy combined with task-specific training (FEST+TST)
- Delayed FEST + TST (Experimental): Participants will receive FEST+TST at 6 to 9 months from SCI onset.
  Interventions: Other: FES Therapy combined with task-specific training (FEST+TST)

INTERVENTIONS:
Other: FES Therapy combined with task-specific training (FEST+TST) — The FEST+TST protocol consists of a 1-hour session, 3 to 5 days a week, for up to 12 weeks (40 sessions total) in addition to conventional occupational and physical therapies according to the standard of care.

SUMMARY:
The purpose of this study is to investigate whether the timing of delivery of functional electrical stimulation therapy in combination with task-specific training (FEST+TST) following spinal cord injury (SCI) influences functional and neurological recovery.

ELIGIBILITY:
Inclusion Criteria:

• Subacute stage (<3 months) after traumatic, motor incomplete (AIS C or D), cervical SCI

Exclusion Criteria:

* Contraindications for neurophysiological tests
* Contraindications for FEST
* Medical conditions that can limit treatment protocols
* Other neurological diseases (i.e. peripheral neuropathies)
* Significant persisting mental illness;
* Learning disabilities;
* Substance abuse over 6 months prior to recruitment;
* Hearing and visual deficits sufficient to affect test performance;
* Contraindication to MRI scanning

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Spinal Cord Independence Measure (SCIM) | Change from baseline SCIM at 3 & 6 months
  Self-care SCIM subscore (0-20) and total SCIM score (0-100) will be used to assess the degree of disability for individuals with SCI with respect to activities of daily living; higher scores reflect greater degree of functional independence
American Spinal Injury Association (ASIA) Upper-Extremity Motor Score (UEMS) | Change from baseline ASIA UEMS score at 3 & 6 months (ASIA UEMS varies from 0 [complete tetraplegia) to 50 [normal])
  International Standards for Neurological Classification of SCI (ISNCSCI) motor and sensory subscores will be used to evaluate degree of impairment.
ASIA Upper-Extremity Sensory Score (UESS) | Change from baseline ASIA UESS score at 3 & 6 months (ASIA UEMS varies from 0 [complete paralysis) to 50 [normal])
  International Standards for Neurological Classification of SCI (ISNCSCI) motor and sensory subscores will be used to evaluate degree of impairment.
Graded Redefined Assessment of Strength Sensibility and Prehension (GRASSP) | Change from baseline GRASSP score at 3 & 6 months (GRASSP score varies from o (complete paralysis) to 148 [normal])
  The GRASSP is a clinical measure used to evaluate upper limb impairment following SCI across 3 domains: strength, sensation, and prehension.

SECONDARY OUTCOMES:
Needle Electromyography | Change in baseline EMG activity at 3 & 6 months
  Disposable monopolar needles will be used to record the insertional activity, spontaneous activity (at rest) and motor unit action potentials (MUAPs) in selected distal muscles (i.e. abductor pollicis brevis and first dorsal interosseous muscles) and proximal muscles (i.e. pronator teres and flexor carpi ulnaris muscles) that are innervated by median and ulnar nerves, respectively, in the dominant (or weaker) upper extremity of each participant.
Repetitive Nerve Stimulation | Change in baseline neuromuscular junction transmission at 3 & 6 months
  Stimulation of the median nerve (and ulnar nerve) in the dominant (or weaker) upper extremity of each individual will be applied using a bar electrode with the responses recorded in the abductor pollicis brevis (APB) muscle (and first dorsal interosseous muscle).
Nerve Conduction Studies | Change in baseline nerve conduction at 3 & 6 months
  Supramaximal stimulation will be applied to the dominant (or weaker) upper extremity of each participant to determine the amplitude, distal latency and conduction velocity from the median and ulnar motor responses.
F-Wave | Change in baseline F-wave amplitude at 3 & 6 months
  Percutaneous supramaximal stimulation will be applied distally to the median nerve (and ulnar nerve) in the dominant (or weaker) upper extremity of each individual with responses recorded from the abductor pollicis brevis muscle (and abductor digiti minimi muscle).
H-Reflex | Change in baseline H-reflex amplitude at 3 & 6 months
  Percutaneous stimulation will be applied to the median nerve of the dominant (or weaker) upper extremity of each individual with responses recorded from the flexor carpi radialis (FCR) muscle using surface electrodes.
Somatosensory Evoked Potentials (SSEPs) | Change in baseline SSEPs at 3 & 6 months
  Electrical stimulation will be applied to the median nerve (and ulnar nerve) in the distal portion of the dominant (or weaker) upper extremity. Recordings will be obtained from the contralateral C3/C4-Fz sites (based in the international 10/20 system) using surface electrodes.
Motor Evoked Potentials (MEPs) | Change in baseline MEPs at 3 & 6 months
  Transcranial magnetic stimulation (TMS) will be used to evoke MEPs in the abductor pollicis brevis muscle (and first dorsal interosseous muscle) of the dominant (or weaker) upper extremity with the coil positioned over the contralateral motor cortex.
Functional Magnetic Resonance Imaging (fMRI) | Change in baseline functional connectivity at 3 & 6 months
  Functional connectivity changes in the motor and somatosensory cortices and pathways will be examined using resting-state fMRI.
Laboratorial Assessments (BDNF) | Change in baseline BDNF at 3 & 6 months
  Blood will be drawn to quantify the presence of brain derived neurotrophic factor [BDNF] in the blood.
Laboratorial Assessments (NTF-3) | Change in baseline NTF-3 at 3 & 6 months
  Blood will be drawn to quantify the presence of neurotrophic factor 3 [NTF-3] in the blood.

CONTACTS AND LOCATIONS:
Overall Officials: Julio Furlan, MD, PhD, Principal Investigator — KITE, Toronto Rehab-University Health Network
Locations (1):
- Lyndhurst Centre, KITE - TRI UHN, Toronto, Ontario, Canada